CLINICAL TRIAL: NCT05525052
Title: Percutaneous Trans-facet Screw Fixation Under CT-scan Guidance for Remaining Symptoms at a Distance of Previous Spinal Surgery: a New Treatment
Brief Title: Percutaneous Trans-facet Screw Fixation Under CT-scan Guidance for Remaining Symptoms at a Distance of Previous Spinal Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22-IMAGERIE-02
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Spinal Stenosis; Spinal Disease; Zygapophyseal Joint Arthritis; Joint Instability; Arthrodesis; Laminectomy; Post Laminectomy Syndrome
MeSH Terms: conditions — Spinal Stenosis; Spinal Diseases; Joint Instability; Ankylosis; post laminectomy syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Patients having a history of spinal surgery such as laminectomy and/or classic surgical arthrodesis, and subsequent focal spinal, treated by transfacet arthrodesis under CT scan guidance
  Interventions: Other: Trans-Facet fixation

INTERVENTIONS:
Other: Trans-Facet fixation — Trans-facet fixation (TFF) under local anesthesia and double fluoroscopic and CT guidance is a minimally invasive technique involving the placement of screws through the posterior facet joints, improving spinal stability.

SUMMARY:
Background : Segmental spinal instability after a laminectomy, and adjacent segment disease (ASD) at after an arthrodesis, are well-known concerns in spinal surgery, which may require re-interventions, usually by surgical arthrodesis, posing the problem of a new heavy intervention under general anesthesia, in often fragile patients.

Trans-facet fixation (TFF) under local anesthesia and double fluoroscopic and CT guidance is a minimally invasive technique involving the placement of screws through the posterior facet joints, improving spinal stability.

Purpose : The aim of our study is to evaluate the efficacy, in terms of pain reduction (VAS) and improvement of daily activities (ODI), of TFF under CT scan guidance in the context of low back pain and/or radiculalgia related to focal instability secondary to laminectomy or ASD.

Methods : TFF were performed in 24 patients having a history of spinal surgery such as laminectomy and/or classic surgical arthrodesis and remaining symptomatic, at Nice University Hospital between 2017 and 2021 Pre- and postoperative pain and disability levels were measured using the visual analogue scale (VAS) and the Oswestry Disability Index (ODI), collected prospectively at systematic 6-month and 1-year follow-up visits. Long term evolution were assessed by phone consultation.

ELIGIBILITY:
Inclusion criterias : - Patients treated at Nice University Hospital between 2017 and 2021 by transfacet arthrodesis,

* History of spinal surgery ( laminectomy and/or classic arthrodesis) - Clinical signs of subsequent instability(low back pain and/or radiculopathy).
* MRI or scintigraphy signs of instability or ASD :
* Spondylolisthesis appeared or increased on successive exams
* Facet dislocation
* Subchondral bone changes of the vertebral endplates (Modic 1)
* Insufficient improvment after epidural and posterior joint corticosteroid infiltrations

Ages: 49 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated at Nice University Hospital between 2017 and 2021 by transfacet arthrodesis, with history of spinal surgery ( laminectomy and/or classic arthrodesis), andsigns of subsequent instability.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) of pain and Oswestry Disability Index (ODI) | 6 months
  Pre- and postoperative pain were measured using the visual analogue scale (VAS), from 0 (no pain) to 10 (maximal pain) collected prospectively at systematic 6-month visit.

SECONDARY OUTCOMES:
pain | From 6 months (systematic consultation) to 4 yours (phone consultation)
  Pre- and postoperative pain and disability levels were measured using the visual analogue scale (VAS)', from 0 (no pain) to 10 (maximal pain)collected prospectively at systematic 1-year follow-up visits. Long term evolution were assessed by phone consultation
Disability | From 6 months (systematic consultation) to 4 yours (phone consultation)
  Pre- and postoperative disability were measured using the Oswestry Disability Index (ODI), from 0 to 100, collected prospectively at systematic 6-months and 1-year follow-up visits. Long term evolution were assessed by phone consultation
Severe intraoperative and postoperative complications | From 6 months (systematic consultation) to 4 yours (phone consultation)
  death , hemorrhage or infection requiring intensive care, post-operative neurological deficit
Need for further interventions afterward the procedure | From 6 months (systematic consultation) to 4 yours (phone consultation)
  need for another surgery
Mean procedure time | At inclusion
  the mean time of procedures in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Vincent SALA, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France